CLINICAL TRIAL: NCT02624271
Title: Non Invasive Diagnosis of Gastric Precancerous Lesions by GastroPanel Blood Test in Patients With Increased Gastric Cancer Risk : a French Multicenter Study
Brief Title: Diagnosis of Gastric Precancerous Lesions by a Blood Test GastroPanel in Patients With Increased Gastric Cancer Risk
Acronym: GASTRO-PRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC14_0371
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer; Gastric Precancerous Lesions
Keywords: gastric cancer; gastric precancerous lesions; blood test
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GastroPanel (Experimental): GastroPanel test on blood samples
  Interventions: Other: blood samples analysis

INTERVENTIONS:
Other: blood samples analysis — Analyze blood samples with GastroPanel test to detect gastric precancerous lesions.

SUMMARY:
Despite the declining incidence, gastric cancer (GC) remains the second leading cause of cancer death worldwide. In France, it is the second digestive cancer with 7,000 new cases per year. It is now well demonstrated that patients with H. pylori infection, atrophic gastritis and intestinal metaplasia, have a high risk of developing GC. It is therefore important to detect these pre-neoplastic lesions at an early stage to improve patients prognosis.

Thus, the aim of this project is to investigate the possible screening of gastric precancerous lesions by a blood test (GastroPanel®) in France, in patients with oesophagogastroduodenoscopy (EGD) prescription.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing oesophagogastroduodenoscopy (EGD) according to usual care
* Patients with increased risk of gastric cancer (at least one of the following criteria):

  * age > 50 years,
  * family cases of gastric cancer,
  * known precancerous lesions,
  * Biermer disease,
  * H. Pylori infection,
  * genetic predisposition (ex: Lynch syndrome),
  * MALT lymphoma,
  * dyspepsia.
* Subjects affiliated with an appropriate social security system

Exclusion Criteria:

* Subjects with known active cancer
* Pregnancy
* Patients receiving proton-pump inhibitors
* Conditions that may interfere with the study objectives according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity of GastroPanel blood test | One assessment at baseline
  The pepsinogen I (PGI) level measure will be compared with the gold standard method (anatomopathological examination of gastric biopsy). Results will be expressed in accordance with Sydney system. Patients will be classified as ill if PGI<30µg/l, healthy if PGI >=30µg/l. The sensitivity of GastroPanel test will be calculated with their 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: MATYSIAK BUDNIK Tamara, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France